CLINICAL TRIAL: NCT04328688
Title: Clindamycin - Trimethoprim/Sulfamethoxazole for Pneumocystis Jiroveci Pneumonia After Solid Organ Transplantation Population (CTSTOP)
Brief Title: Clindamycin-trimethoprim/Sulfamethoxazole for PCP After Solid Organ Transplantation Population.
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CTSTOP
Record Dates: First submitted 2020-01-02; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pneumocystis Jirovecii Pneumonia; Solid Organ Transplantation
Keywords: TMP-SMX; clindamycin; oxygenation index; adverse reactions
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PCP is one of the common opportunistic infections in patients with HIV and non-HIV-associated immunodeficiency.With the increasing number of solid organ transplantation, how to effectively treat severe PCP after solid organ transplantation has become an urgent problem to be solved.In general, Atovaquone, Dapsone, and Clindamycin-primaquine can be used as second-line alternatives when TMP-SMX fails to treat HIV-PCP. Therefore, the objective of this study is to preliminarily investigate the safety and efficacy of low-dose TMP-SMX combined with clindamycin (CT regimen) for the treatment of severe PCP after solid organ transplantation.

DETAILED DESCRIPTION:
PCP is one of the common opportunistic infections in patients with HIV and non-HIV-associated immunodeficiency.With the increasing number of solid organ transplantation, how to effectively treat severe PCP after solid organ transplantation has become an urgent problem to be solved.In general, Atovaquone, Dapsone, and Clindamycin-primaquine can be used as second-line alternatives when TMP-SMX fails to treat HIV-PCP. More and more studies suggest that clindamycin-based alternatives play an increasingly important role in treating of PCP. Therefore, the objective of this study is to preliminarily investigate the safety and efficacy of low-dose TMP-SMX combined with clindamycin (CT regimen) for the treatment of severe PCP after solid organ transplantation.

ELIGIBILITY:
Inclusion Criteria:

* PJP after solid organ transplantation.

Exclusion Criteria:

* renal failure,heart failure,tumor recurrence

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A. the clinical manifestations are fever, shortness of breath, dry cough ,respiratory distress B. Chest CT showed manifested by fine, bilateral, perihilar, diffuse infiltrates , an interstitial alveolar butterfly pattern C. Bronchoalveolar lavage was sent for next generation sequencing (NGS)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
oxygenation index | through study completion, an average of 20 days
  PaO2/FiO2
length of ICU stay | through study completion, an average of 20 days
  Total length of stay in ICU

SECONDARY OUTCOMES:
adverse reactions of drugs | through study completion, an average of 20 days
  Rash，Anorexia，Decreased white blood cell count，Anemia，Decreased platelet count，Increased TB，Increased creatinine，Hyperkalemia

CONTACTS AND LOCATIONS:
Locations (1):
- Ju Minjie, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Gu ZY, Liu WJ, Huang DL, Liu YJ, He HY, Yang C, Liu YM, Xu M, Rong RM, Zhu DM, Luo Z, Ju MJ. Preliminary Study on the Combination Effect of Clindamycin and Low Dose Trimethoprim-Sulfamethoxazole on Severe Pneumocystis Pneumonia After Renal Transplantation. Front Med (Lausanne). 2022 May 6;9:827850. doi: 10.3389/fmed.2022.827850. eCollection 2022. PMID 35602475